CLINICAL TRIAL: NCT03177629
Title: Efficacy of Helicobacter Pylori Eradication for the Treatment of Chronic or Persistent Immune Thrombocytopenic Purpura Patients With Moderate Thrombocytopenia: Multicenter Prospective Randomized Phase 3 Study
Brief Title: H. Pylori Eradication for Moderate ITP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Hallym University Medical Center (Other)
Responsible Party: Principal Investigator, Soo-Mee Bang, Professor, Department of Internal Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSH_ITP1701
Record Dates: First submitted 2017-05-29; First posted 2017-06-06 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Immune Thrombocytopenic Purpura; Helicobacter Pylori; Immune Thrombocytopenia
Keywords: Immune Thrombocytopenic Purpura; Helicobacter pylori
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Intervention Model Description: treatment group vs control group Patients in treatment group will be treated with antibiotics for H. pylori eradication at visit 1.
  Control group has 2 stage. Fot the 1st stage (for 3 months), the patient will be observed without any treatment. And at visit 4, at 2nd stage, they will be treated with the same regimen for H. pylori eradication.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment arm: H. pylori eradication (Experimental): treatment arm: H. pylori eradication at visit 1(0 month)
  Interventions: Drug: treatment : H. pylori eradication
- Control arm -1st stage (No Intervention): At visit 1(0 month) no intervention, observation only from visit 1 to visit 3
- Control arm - 2nd stage (Active Comparator): Same patients group with control arm 1st stage. After observation for 3 months during stage 1, the patients of control arm will be treated with same regimen for H. pylori eradication at visit 4 (2nd stage).
  Interventions: Drug: treatment : H. pylori eradication

INTERVENTIONS:
Drug: treatment : H. pylori eradication — treatment: H. pylori eradication (pantoprazole, amoxicillin, clarithromycin, metronidazole) to treatment group at visit 1 and to control group 2nd stage at visit 4.
  Day 1-5: pantoprazole 40mg bid, amoxicillin 1000mg bid, PO Day 6 - 10: pantoprazole 40mg bid, clarithromycin 500mg bid, metronidazole 500mg tid, PO
  Arms: Control arm - 2nd stage; Treatment arm: H. pylori eradication

SUMMARY:
The purpose of this study is to determine the efficacy of H. pylori eradication for the treatment of chronic or persistent immune thrombocytopenic purpura (ITP) patients with moderate thrombocytopenia. This is a multi-center, open label, prospective randomized phase IIl study.

DETAILED DESCRIPTION:
Current treatment guideline of ITP recommends corticosteroid as the first line treatment when patient has active bleeding or less than 30×10^9/L of platelet, because of side effect and cost issues. Since the first case report by Italian study, several investigators have reported that secondary immune thrombocytopenia (ITP) can occur in patients with Helicobacter pylori (H. pylori) infection. We already reported the efficacy of H. pylori eradication in moderate ITP patients with phase II study (Annals Hematology 2015:94:739-46). To improve the evidence of this strategy for the treatment of moderate ITP, we plan to start this multi-center, open label, prospective randomized phase 3 study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 19 years
* Persistent or chronic ITP patients defined by international working group
* 30 X 10^9/L ≤ platelet level ≤ 80 X 10^9/L
* H. pylori infection should be confirmed by at least one of tests: urea breath test (UBT), CLO, stool H. pylori Ag, H. pylori in gastric tissue (reported by a trained pathologist)
* No history of any ITP treatment for the past 3 months
* No previous history of H. pylori eradication treatment
* Patients who voluntarily participate in this study and with informed consents

Exclusion Criteria:

* patients who have any cause of thrombocytopenia such as HIV, HCV infection, lymphoproliferative disease, malignant neoplasm, liver disease, definite SLE and other autoimmune diseases, drugs, MDS and leukemia
* uncontrolled hypothyroidism or hyperthyroidism
* active bleeding for the past 3 months or history of hemorrhagic gastric ulcer or brain hemorrhage
* active infection
* patients who are taking anticoagulant or aspirin
* patients with penicillin allergy or side effects of macrolide
* patients who are taking mizolastine, terfenadine, cisapride, pimozide, astemizole, ergot alkaloid and its derivatives (ergotamine and dihydroergotamine), bepridil or atazanavir
* patients who have known allergy or severe side effect on study drugs
* pregnant or lactating women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-05-23 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR: complete response + response rate) of platelets | visit 4 (3 months after randomization)
  1. ORR between treatment group with UBT (-) and control group with stage 1
  2. International working group criteria for ITP treatment response will be used for ORR definition

SECONDARY OUTCOMES:
ORR between treatment group and control group with stage 1 | visit 4 (3 months after randomization)
  all patients in the treatment group (with UBT (+) or UBT (-) patients)
ORR of control group with stage 2 | At visit 5 (6 months after randomization)
  patients in the control group with stage 2 with UBT (-)
ORR after H. pylori eradication in all patients who were treated and UBT (-) | 3 months after H. pylori eradication
  UBT (-) patients in treatment group and control group with stage 2
Time to response | from initiation date of study drugs to the date of R or CR (assessed up to 6 months)
  from initiation date of study drugs to the date of R or CR in treatment group
Response duration | from the date of R or CR to the date of loss of R or CR / or till last f/u date, whichever came first (assessed up to 6 months)
  from the date of R or CR to the date of loss of R or CR / or till last f/u date in treatment group
H. pylori eradication rate | at vist 4 (3 months after randomization) after drug treatment
  defined by UBT (-)
drug toxicity and compliance | At visit 2, 3, 4, 5 (1, 2, 3, 6 months after randomization, respectively) for treatment group, at visit 5 (6 months after randomization) for control group stage 2
  NCI CTCAE v4.0 for safety measurement, 85% of taking medicine for criteria of compliance
QoL | At visit 1(Day 1 of study drug medication) & vist 4 (3 months after randomization)
  within & between group after H. pylori eradication, FACIT-F, FACIT-Th6
platelet level at randomization | 3 months after H. pylori eradication
  comparison of platelet level at randomization between treatment responder and non-responder of H. pylori eradication
ITP duration before randomization | 3 months after H. pylori eradication
  comparison of ITP duration before randomization between treatment responder and non-responder of H. pylori eradication

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Me Bang, M.D., Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim H, Lee WS, Lee KH, Bae SH, Kim MK, Joo YD, Zang DY, Jo JC, Lee SM, Lee JH, Lee JH, Kim DY, Ryoo HM, Hyun MS, Kim HJ; CoOperative Study Group A for Hematology (COSAH). Efficacy of Helicobacter pylori eradication for the 1st line treatment of immune thrombocytopenia patients with moderate thrombocytopenia. Ann Hematol. 2015 May;94(5):739-46. doi: 10.1007/s00277-014-2268-9. Epub 2014 Dec 13. PMID 25501820
- [Derived] Han B, Kim HJ, Yhim HY, Oh D, Bae SH, Shin HJ, Lee WS, Kwon J, Lee JO, Kim HJ, Bang SM. Sequential eradication of Helicobacter pylori as a treatment for immune thrombocytopenia in patients with moderate thrombocytopenia: a multicenter prospective randomized phase 3 study. Ann Hematol. 2022 Jul;101(7):1435-1445. doi: 10.1007/s00277-022-04782-2. Epub 2022 May 28. PMID 35643952